CLINICAL TRIAL: NCT01887548
Title: Personality Traits and Its Impact on Quality of Life and Clinical Outcome Evaluation in Patients With Crohn's Disease
Brief Title: Personality Traits and Its Impact on Quality of Life and Clinical Outcome Evaluation in Crohn's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Vice president of department of surgery, Jinling Hospital, Jinling Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20130618
Record Dates: First submitted 2013-06-19; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; inflammatory bowel disease; quality of life; personality; neuroticism
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active CD (Experimental): Patients whose CDAI score >150 points would be enrolled in this group.
  Interventions: Other: Personality Traits Questionnaires
- Quiescent CD (Active Comparator): Patients whose CDAI score ≤150 points would be enrolled in this group.
  Interventions: Other: Personality Traits Questionnaires

INTERVENTIONS:
Other: Personality Traits Questionnaires — Patients are required to fill out several personality traits questionnaires. The following personality traits scores would be collected: IBDQ, IBDQ-Emotional function score, IBDQ-Social function score, IBDQ-Bowel function score, IBDQ-Systemic symptom score, Neuroticism score, Lie (social conformity/desirability) score, Hospital anxiety score, Hospital depression score, Buss-Perry score, PA (physical aggression) score, VA (verbal aggression) score, A (anger) score, H (hostility) score.

SUMMARY:
Quality of life is recommended as one of essential parameters to evaluate treatment effect and clinical outcome in patients with Crohn's disease (CD). Recent studies reported that several disease-unrelated variables may affect quality of life in CD patients. This study is dedicated to investigate the influence of various personality traits on quality of life, and whether or not they should be taken into account when evaluating clinical outcomes in patients with CD.

DETAILED DESCRIPTION:
This is a prospective, single-center study.

All enrolled patients are divided into 2 groups:

* Group 1: quiescent CD group (CDAI≤150 points)
* Group 2: active CD group (CDAI>150 points)

All enrolled patients are required to accomplish the following questionnaires at visit:

* Inflammatory Bowel Disease Questionnaire (IBDQ)
* Neuroticism (N) and Lie (L) subscale of the Eysenck Personality Inventory (EPI)
* Hospital Anxiety and Depression Scale (HADS)
* Buss-Perry Aggression (BPA) questionnaire

All questionnaires are translated and validated in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* a definite diagnosis of CD

Exclusion Criteria:

* current or previous mental disorders
* receiving or once received psychotherapy
* presence of major medical conditions (such as necessity of an operation)
* chronic disease history other than inflammatory bowel disease
* unwilling to participate in or cannot accomplish current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
IBDQ | one week
  Inflammatory Bowel Disease Questionnaires (IBDQ) is the most widely used and validated disease-specific instrument, which contains 32 items and assesses four aspects (subscales) of quality of life: emotional function (12 items), social function (5 items), bowel function (10 items) and systemic symptom (5 items).

SECONDARY OUTCOMES:
Eysenck Personality Inventory (EPI) | one week
  To assess neuroticism and social conformity and desirability, the Neuroticism and Lie subscales from the Eysenck Personality Inventory (EPI) were adopt in current study. Twenty-three items are designed to evaluate neuroticism (Neuroticism subscale) and the other 21 items are assigned for social desirability (Lie subscale).
Hospital Anxiety and Depression Scale (HADS) | one week
  The Hospital Anxiety and Depression Scale (HADS) was first developed in 1983 and has been extensively used in subsequent studies to identify the potential anxiety and depression in nonpsychiatric hospitalized patients. This questionnaire includes separated Anxiety and Depression subscales with seven items, respectively.
Buss Perry Aggregation (BPA) questionnaire | one week
  BPA is one of the most popular self-report inventories for the measurement of four different dimensions (anger, hostility, physical aggression and verbal aggression). This 29-item questionnaire is scored with a 5-level scale for each question, contributing to a total score and four subscales of each dimension. A higher score suggests a higher level of aggression feelings.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Jinling Hospital, Nanjing, Jiangsu, China